CLINICAL TRIAL: NCT06138639
Title: A Phase 1/2, Multicenter, Open-Label Study to Investigate the Safety, Tolerability, and Efficacy of a Single Intravenous Dose of SGT-003 in Males With Duchenne Muscular Dystrophy (INSPIRE DUCHENNE)
Brief Title: A Study of SGT-003 Gene Therapy in Duchenne Muscular Dystrophy (INSPIRE DUCHENNE)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Solid Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGT-003-101; 2024-514501-57-00 (EU CTIS Number); 1010251 (Other: UK IRAS ID)
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: DMD; Gene Therapy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Cohort 1: SGT-003 (Experimental): All ambulatory participants from age 4 to < 7 years will receive a single IV infusion of SGT-003 on Day 1.
  Interventions: Genetic: SGT-003
- Cohort 2: SGT-003 (Experimental): All ambulatory participants from age 7 to < 12 years will receive a single IV infusion of SGT-003 on Day 1.
  Interventions: Genetic: SGT-003
- Cohort 3: SGT-003 (Experimental): All participants from age 0 to < 4 years will receive a single IV infusion of SGT-003 on Day 1.
  Interventions: Genetic: SGT-003
- Cohort 4: SGT-003 (Experimental): All ambulatory participants from age 12 to < 18 years will receive a single IV infusion of SGT-003 on Day 1.
  Interventions: Genetic: SGT-003
- Cohort 5: SGT-003 (Experimental): All non-ambulatory participants from age 10 to < 18 years will receive a single IV infusion of SGT-003 on Day 1.
  Interventions: Genetic: SGT-003

INTERVENTIONS:
Genetic: SGT-003 — Adeno-associated virus serotype SLB101 containing the human microdystrophin gene (h-µD5)

SUMMARY:
This is a multicenter, open-label, non-randomized study to investigate the safety, tolerability, and efficacy of a single intravenous (IV) infusion of SGT-003 in participants with Duchenne muscular dystrophy. There will be 5 cohorts in this study. Cohort 1 will include participants 4 to < 7 years of age. Cohort 2 will include participants 7 to < 12 years of age. Cohort 3 will include participants 0 to < 4 years of age. Cohort 4 will include participants 12 to < 18 years of age. Cohort 5 will include participants 10 to < 18 years of age. Initiation of participant enrollment in Cohorts 4 and 5 will be subject to the accrual of safety and efficacy data from Cohorts 1-3. All participants will receive SGT-003 and will be enrolled in the study for 5 total years for long-term follow up.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1: 4 to <7 years of age
* Cohort 2: 7 to <12 years of age
* Cohort 3: 0 to < 4 years of age
* Cohort 4: 12 to < 18 years of age
* Cohort 5: 10 to < 18 years of age
* Participant ambulatory status at the time of Screening Part A or Rescreening, as defined by the ability to complete a 10-meter walk/run test in < 30 seconds:

  * Cohorts 1, 2, and 4: Ambulatory
  * Cohort 3: Either ambulatory or non-ambulatory
  * Cohort 5: Non-ambulatory, but having been previously ambulatory by history
* Established clinical diagnosis of DMD and documented dystrophin gene mutation predictive of DMD phenotype confirmed by Sponsor genetic testing. In cases where a genotype may be predictive of residual dystrophin production and/or a clear clinical diagnosis of DMD cannot be made (e.g., due to age), evaluation of dystrophin levels in baseline muscle biopsies may be required to determine eligibility under this criterion.
* Negative for AAV antibodies.
* Steroid regimen:

  * Cohorts 1, 2, 4, and 5: A stable daily oral steroid regimen of at least 0.5 mg/kg/day of prednisone or 0.75 mg/kg/day of deflazacort for ≥12 weeks prior to Screening Part A or Rescreening, allowing for weight-based modifications consistent with clinical practice.
  * Cohort 3: N/A
* Meet 10-meter walk/run time criteria
* Meet time to rise from supine criteria
* Cohort 5: Meet Performance of Upper Limb (PUL) 2.0 criteria
* Participant has body weight: ≤ 90 kg

Exclusion Criteria:

* Treatment with dystrophin modifying drugs within 3 months prior to screening.
* Current or prior treatment with an approved or investigational gene transfer drug.
* Exposure to certain approved or investigational drugs within 3 months prior to screening or 5 half-lives since last administration, whichever is longer.
* Established clinical diagnosis of DMD that is associated with any deletion mutation invariant or variant predicted to not express exons 1 to 11 or, exons 42 to 45, or exons 57 to 69, inclusive, in the DMD gene as documented by a genetic report and confirmed by Sponsor genetic testing.

Other inclusion or exclusion criteria apply.

Ages: 0 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2027-05-06 (Estimated); Study Completion 2031-05-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (AEs) | Day 360
Change from baseline in Microdystrophin Protein Levels | Day 90
  Microdystrophin expression evaluation in muscle biopsies

SECONDARY OUTCOMES:
Change from Baseline of Microdystrophin Tissue Distribution by Immunofluorescence (IF) | Day 90, Day 360
Change from baseline in Microdystrophin Protein Levels | Day 360
  Microdystrophin expression evaluation in muscle biopsies
Change from Baseline in Time to Rise Velocity | Day 360, Day 540
  The Time to rise from supine (TTR) (s) will be captured as part of item 12 of the North Star Ambulatory Assessment (NSAA).
  Assessment of muscle function using a 17-item scale with each item scored from 0 to 2 and a higher score meaning a better outcome. The NSAA total score is defined as the sum of all 17 items, ranging from 0 to 34, with a higher score meaning a better outcome.
Change from baseline in Stride Velocity 95th Centile (SV95C) | Day 360, Day 540
  Assessment of peak ambulatory performance captured by wearable activity monitoring device.
Change from baseline in 10-meter walk/run velocity | Day 360, Day 540
  The 10MWR (s) will be captured as part of item 17 of the NSAA. Assessment of muscle function using a 17-item scale with each item scored from 0 to 2 and a higher score meaning a better outcome. The NSAA total score is defined as the sum of all 17 items, ranging from 0 to 34, with a higher score meaning a better outcome.
Change from baseline in 4-stair climb velocity | Day 360, Day 540
Change from baseline in North Star Ambulatory Assessment (NSAA) total score | Day 360, Day 540
  Assessment of muscle function using a 17-item scale with each item scored from 0 to 2 and a higher score meaning a better outcome. The NSAA total score is defined as the sum of all 17 items, ranging from 0 to 34, with a higher score meaning a better outcome.
Change from baseline in 6-minute walk test (6MWT) distance | Day 360, Day 540
Number of Participants with Clinically Significant Abnormalities in Laboratory Parameters | Through Day 360 and Day 540
Number of Participants with Clinically Significant Abnormalities in Vital Signs | Through Day 360 and Day 540
Number of Participants with Clinically Significant Abnormalities in Physical Examinations | Through Day 360 and Day 540
Number of Participants with Clinically Significant Abnormalities in Electrocardiogram (ECG) or Echocardiography (ECHO) | Through Day 360 and Day 540

CONTACTS AND LOCATIONS:
Overall Officials: Solid Bio Clinical Trials, Study Director — Solid Biosciences
Locations (15):
- United States (12):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of California, Los Angeles Medical Center, Los Angeles, California
  - University of California, Davis, Sacramento, California
  - University of California, San Diego, California
  - Rare Disease Research, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Washington University in St. Louis, St Louis, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Sciences University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
- The Hospital for Sick Children, Toronto, Ontario, Canada
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy
- Great Ormond Street Hospital, London, United Kingdom